CLINICAL TRIAL: NCT05189132
Title: Periodonitis and Alzheimer's Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Lisbon (Other)
Responsible Party: Principal Investigator, Vanessa Rocha Rodrigues, Principal Investigator, University of Lisbon
Other Study IDs: University Lisbon
Record Dates: First submitted 2021-12-26; First posted 2022-01-12 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Alzheimer Disease; Periodontitis
Keywords: Alzheimer Disease; Periodontitis
MeSH Terms: conditions — Alzheimer Disease; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test Group: Adult patients diagnosed with Alzheimer's disease
  Interventions: Diagnostic Test: Periodontal Diagnosis; Diagnostic Test: Microbiological analysis; Diagnostic Test: Inflammatory mediators
- Control Group: The control group will consist of patients who attend consultations at the Faculty of Dentistry of the University of Lisbon, matched for age, gender and other confounding factors, such as smoking and systemic diseases (diabetes).
  Interventions: Diagnostic Test: Periodontal Diagnosis; Diagnostic Test: Microbiological analysis; Diagnostic Test: Inflammatory mediators

INTERVENTIONS:
Diagnostic Test: Periodontal Diagnosis — All participants, in the test group and in the control group, will undergo an initial periodontal evaluation. The clinical evaluation will always be carried out by the same examiner, the author of the study, in order to guarantee calibrated observations. During data collection, intra-observer calibration will be performed, as recommended by the WHO (WHO, 1993), in order to minimize diagnostic variability and verify agreement
Diagnostic Test: Microbiological analysis — Microbiological analysis will be performed using a sample of subgingival bacterial plaque. The sample will be collected at the tooth and at the location with the highest probing depth values in each quadrant.
  A sterilized paper tip from the microbiological kit will be introduced to the bottom of the bag, with the aid of tweezers, remaining in the same position for 10 seconds. After collecting the sample, the paper tip will be placed in an individual transfer tube, properly identified. Afterwards, the sample will be sent to the laboratory, where a polymerase chain reaction (PCR) test is performed to identify the following bacteria - A. actinomycetemcomitans, T. forsythia, T. denticola, P. gingivalis, P. intermedia and F. nucleatum.
Diagnostic Test: Inflammatory mediators — The evaluation of inflammatory mediators will be performed with the aid of an absorbent paper strip, which is placed inside the periodontal pocket, for about 30 seconds. The sample will be taken from the tooth that has the highest probing depth values.
  The collected sample will be placed and stored in an individual transfer tube properly identified and in accordance with the laboratory's instructions. Afterwards, the sample will be sent to the laboratory, where the ELISA test is performed to quantify the following inflammatory mediators - IL-1β, IL-6 and TNF-α.

SUMMARY:
The main objective of this study is to assess whether Periodontal Disease is more prevalent in adult patients diagnosed with Alzheimer's Disease compared to adult patients without Alzheimer's Disease.

The secondary objective is to describe and characterize the microbiological and biochemical profile of adult patients diagnosed with Alzheimer's Disease and compare with adult patients without Alzheimer's Disease.

DETAILED DESCRIPTION:
To assess the possible association of Periodontal Disease with Alzheimer's Disease, I propose to carry out an observational, paired and cross-sectional study.

It will be evaluated whether adult patients diagnosed with Alzheimer's Disease have a higher prevalence of Periodontal Disease when compared to adult patients without Alzheimer's Disease.

As well, it will be evaluated whether adult patients with different stages of Alzheimer's disease have different stages of severity of Periodontitis.

The study sample will be obtained from the Associação Portuguesa de Alzheimer, in the Lisbon region, consisting of adult patients diagnosed with Alzheimer's Disease (test group).

The control group sample will consist of patients who attend consultations at the Faculty of Dental Medicine, University of Lisbon, matched for age, gender and other confounding factors, such as tobacco and systemic diseases (diabetes).

ELIGIBILITY:
Inclusion Criteria:

Will be included in the study all individuals who attend the Portuguese Alzheimer's Association, diagnosed with Alzheimer's Disease, who:

1. have voluntarily given their consent to participate;
2. due to cognitive or functional disability, they were unable to give free and informed consent, but they had this consent given by their representative
3. individuals who have participated in the cognitive assessment (only for the test group)

Exclusion Criteria:

* a) refused oral observation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: It will be evaluated whether adult patients diagnosed with Alzheimer's Disease have a higher prevalence of Periodontal Disease when compared to adult patients without Alzheimer's Disease.
  As well, it will be evaluated whether adult patients with different stages of Alzheimer's disease have different stages of severity of Periodontitis.
  The study sample will be obtained from the Associação Portuguesa de Alzheimer, in the Lisbon region, consisting of adult patients diagnosed with Alzheimer's Disease (test group).
  The control group sample will consist of patients who attend consultations at the Faculty of Dental Medicine, University of Lisbon, matched for age, gender and other confounding factors, such as tobacco and systemic diseases (diabetes).
Sampling Method: Non-Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Probing depth | Basline
  The probing depth corresponds to the distance from the gingival margin to the bottom of the sulcus or periodontal pocket. Probing depth measurement will be performed at six locations per tooth, three locations per buccal and three locations per lingual/palatal
Clinical attachment level | Basline
  The clinical insertion level corresponds to the distance from an enamel-cementary junction (JAC) to the bottom of the pocket.
  * In cases where there is gingival recession, the insertion level is complete through the sum of the probing depth value and the gingival recession value (distance from the gingival margin to the JAC).
  * In cases where the gingival margin coincides with the JAC, the insertion level value is the same as the probing depth.
  * If there is a pseudo-pocket, characterized by an increase in gingival volume in the coronal direction, the insertion level value will be the result of subtracting the probing depth value and the distance from the gingival margin to the JAC.
Plaque index | Basline
  For the evaluation of the plaque index (PI), the PI developed by the authors Ainamo and Bay, in 1975, will be used. It is a dichotomous index, which assesses the presence or absence of bacterial plaque in the cervical area of the tooth in four locations, three locations by vestibular and one location by palatine
Bleeding on probing | Basline
  Bleeding on probing is assessed by looking at bleeding points after periodontal probing. It will be evaluated in six locations per tooth, three locations per buccal and three locations per lingual/palatal. A red circle is placed around the sounding depth value (Lang 1986 and 1990).
Gingival Recessions | Basline
  Gingival recession will be evaluated in millimeters and is obtained by the distance from the gingival margin to the JAC. It will be evaluated in six locations per tooth, three locations per buccal and three locations per lingual/palatal
Mobility | Basline
  Mobility will be assessed with the handle of two instruments (probe and mirror), pushing the tooth in the buccolingual and occlusal-apical directions.
  The classification proposed by Miller in 1950 will be used, which is divided into: Mobility 0: physiological (0mm to 0.2mm);
  * Mobility I: < 1mm in the horizontal direction;
  * Mobility II: > 1mm in the horizontal direction;
  * Mobility III: horizontal and vertical mobility.
Furcation | Basline
  The presence of furcation lesions will be evaluated using the Nabers probe. Will be used in the 1975 classification of Hamp
  * Grade 1 - Loss of horizontal insertion tissue less than 3mm
  * Grade 2- Loss of horizontal insertion tissue greater than 3mm, but the probe does not it passes from one side to the other.
  * Grade 3- Loss of horizontal insertion tissue greater than 3mm and the probe passes from side to side

SECONDARY OUTCOMES:
Microbiological analysis | Basline
  Microbiological analysis will be performed using a sample of subgingival bacterial plaque. The sample will be collected at the tooth and at the location with the highest probing depth values in each quadrant.
  A sterilized paper tip from the microbiological kit will be introduced to the bottom of the bag, with the aid of tweezers, remaining in the same position for 10 seconds. After collecting the sample, the paper tip will be placed in an individual transfer tube, properly identified. Afterwards, the sample will be sent to the laboratory, where a polymerase chain reaction (PCR) test is performed to identify the following bacteria - A. actinomycetemcomitans, T. forsythia, T. denticola, P. gingivalis, P. intermedia and F. nucleatum.
Inflammatory Mediators | Basline
  The evaluation of inflammatory mediators will be performed with the aid of an absorbent paper strip, which is placed inside the periodontal pocket, for about 30 seconds. The sample will be taken from the tooth that has the highest probing depth values.
  The collected sample will be placed and stored in an individual transfer tube properly identified and in accordance with the laboratory's instructions. Afterwards, the sample will be sent to the laboratory, where the ELISA test is performed to quantify the following inflammatory mediators - IL-1β, IL-6 and TNF-α

OTHER OUTCOMES:
Cognitive Assessment | Basline
  Cognitive assessment will be performed by neurologists from the Portuguese Alzheimer's Association.
  Periodontal diagnosis will be performed, through clinical evaluation, to patients with and without Alzheimer's Disease. The Classification of Periodontal and Peri-implant Diseases and Conditions proposed by the American Association of Periodontology (AAP) and the European Federation of Periodontology (EFP) will be used to determine the prevalence of periodontal disease.
  To assess whether adult patients with different stages of Alzheimer's disease have different stages of severity of Periodontitis (I, II, III and IV), in addition to a periodontal evaluation, it is also evaluated through cognitive tests, at which stage of the disease Alzheimer's patient is found.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Rocha Rodrigues, Dr, Principal Investigator — University of Lisbon

IPD SHARING:
Plan to Share IPD: Undecided